CLINICAL TRIAL: NCT04332016
Title: Biological Samples Collection From Patients and Caregivers Treated at Bordeaux University Hospital for Asymptomatic and Symptomatic Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) Infection (COVID-19).
Brief Title: COVID-19 Biological Samples Collection
Acronym: COLCOV19-BX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/11
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Infection Viral
Keywords: COVID-19; SARS-CoV-2; coronavirus; biological samples
MeSH Terms: conditions — Virus Diseases; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Sample Upper respiratory sampling Urine and stool collection Post mortem biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infected patients
  Interventions: Other: biological samples collection

INTERVENTIONS:
Other: biological samples collection — collection of whole blood samples, urine and stool samples, upper respiratory samples, post-mortem biopsies

SUMMARY:
The coronavirus disease 2019 (COVID-19) outbreak is now considered as a public health emergency of international concern by the World Health Organization.

In the context of the health emergency, research on the pathogen (the SARS-CoV-2 coronavirus), the disease and the therapeutic care is being organized. Research projects require the use of biological samples. This study aims at setting up a collection of biological samples intended for application projects in any discipline.

The main objective of the study is to collect, process and store biological samples from patients and caregivers infected with SARS-CoV-2 (COVID-19) at the biological ressources center of the Bordeaux University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients / caregivers treated at Bordeaux University Hospital for asymptomatic or symptomatic infection by SARS -CoV-2
* men and women, adults and minors as well as pregnant or breastfeeding women
* patients who died following infection with SARS-CoV-2 (specific criterion for post-mortem biopsies)
* Be affiliated with or beneficiary of a social security scheme
* Free and informed consent obtained and signed by the patient

Exclusion Criteria:

* Under guardianship or curatorship

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients / caregivers treated at Bordeaux University Hospital for asymptomatic or symptomatic infection by SARS -CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
COVID-19 desease description | Inclusion visit (Day 1)
  From blood samples: protein levels, whole genome sequence, transcriptomic analysis data.
  From upper respiratory samples: protein levels, virus transcriptomic analysis data.
  From stool: microbiota analysis data.
  From urine: protein level.
COVID-19 desease description | Day 30 to 90
  From blood samples: protein levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia G, Labrouche-Colomer S, Duvignaud A, Clequin E, Dussiau C, Tregouet DA, Malvy D, Prevel R, Zouine A, Pellegrin I, Goret J, Mamani-Matsuda M, Dewitte A, James C. Impaired balance between neutrophil extracellular trap formation and degradation by DNases in COVID-19 disease. J Transl Med. 2024 Mar 7;22(1):246. doi: 10.1186/s12967-024-05044-7. PMID 38454482